CLINICAL TRIAL: NCT05400629
Title: Effects of a 12-week Strength Training Program in Women With Myotonic Dystrophy Type 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Rare Disease Foundation (Unknown)
Responsible Party: Principal Investigator, Élise Duchesne, Professor Investigator, Université de Sherbrooke
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-005
Record Dates: First submitted 2022-05-24; First posted 2022-06-01 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Myotonic Dystrophy 1
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Intervention Model Description: Participants will complete a 12-week strength training program and return to their normal activities for the following 6 months after the end of the training program.
Masking Description: Most outcomes will not be mask, however the outcome assessor will be mask for all muscle biopsy analysis: while analysing the muscle biopsy outcomes, the outcome assessor will not know if it was from baseline or from after the training program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training program (Experimental): 12-week strength training program of the lower limbs consisting of 5 different exercises: Leg extension, leg press, hip abduction, squat and plantar flexion. All exercises will be perform between 6 and 8 maximal repetitions.
  Interventions: Other: Training program

INTERVENTIONS:
Other: Training program — 12-week strength training program of the lower limbs consisting of 5 different exercises: Leg extension, leg press, hip abduction, squat and plantar flexion. All exercises will be perform between 6 and 8 maximal repetitions.

SUMMARY:
20 women with myotonic dystrophy type 1 (DM1) will complete a 12-week lower-limb strength training program. The training program consist of 3 series of 6 to 8 maximal repetitions of 5 different exercises: Leg extension, leg press, hip abduction, squat and plantar flexion. Training sessions will be closely supervise and take place twice a week. It is hypothesize that the training program will induce muscular hypertrophy despite the genetic defect. The training program should also have positive effects on function. The participants will be evaluated at baseline, week 6, week 12, month 6 and month 9 to quantify the effects of the training program and if these effects will be maintained over time.

ELIGIBILITY:
Inclusion Criteria:

* DM1 diagnosis must be confirmed by genetic analysis;
* Women sex, aged between 30 and 65 years old;
* Be able to walk without assistance;
* Consent of the neurologist must be given to participate in this study;
* Must reside in the Saguenay-Lac-St-Jean region;
* Subjects must be able to give their consent freely and voluntarily.

Exclusion Criteria:

* Patients with any other form of muscular dystrophy are excluded;
* Any contraindication for strenuous exercise or muscle biopsy.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Changes in maximal isometric muscle strength of the knee extensors | At baseline, week 6, week 12, month 3 and month 6
  Changes in maximal isometric muscle strength of the knee extensors measure by quantify muscle testing using a handheld dynamometer

SECONDARY OUTCOMES:
Changes in maximal isometric muscle strength of the knee flexors | At baseline and week 12
  Changes in maximal isometric muscle strength of the knee flexors measure by quantify muscle testing using a handheld dynamometer
Changes in maximal isometric muscle strength of the hip flexors | At baseline and week 12
  Changes in maximal isometric muscle strength of the hip flexors measure by quantify muscle testing using a handheld dynamometer
Changes in maximal isometric muscle strength of the hip extensors | At baseline and week 12
  Changes in maximal isometric muscle strength of the hip extensors measure by quantify muscle testing using a handheld dynamometer
Changes in maximal isometric muscle strength of the hip abductors | At baseline and week 12
  Changes in maximal isometric muscle strength of the hip abductors measure by quantify muscle testing using a handheld dynamometer
Changes in maximal isometric muscle strength of the ankle dorsiflexors | At baseline and week 12
  Changes in maximal isometric muscle strength of the ankle dorsiflexors measure by quantify muscle testing using a handheld dynamometer
Changes in maximal isometric grip strength | At baseline and week 12
  Changes in maximal isometric muscle strength of prehension measure by quantify muscle testing using a hand grip dynamometer
Changes in 1-repetition maximum strength of the leg extension exercise | At baseline, week 6 and week 12
  Changes in 1-repetition maximum strength of the leg extension exercise
Changes in 1-repetition maximum strength of the leg press exercise | At baseline, week 6 and week 12
  Changes in 1-repetition maximum strength of the leg press exercise
Changes in 1-repetition maximum strength of the hip abduction exercise | At baseline, week 6 and week 12
  Changes in 1-repetition maximum strength of the hip abduction exercise
Changes in 1-repetition maximum strength of the squat exercise | At baseline, week 6 and week 12
  Changes in 1-repetition maximum strength of the squat exercise
Changes in comfortable walking speed in the 10-meter walk test | At baseline, week 6, week 12, month 6 and month 9
  Changes in comfortable walking speed in the 10-meter walk test
Changes in maximal walking speed in the 10-meter walk test | At baseline, week 6, week 12, month 6 and month 9
  Changes in maximal walking speed in the 10-meter walk test
Changes in the number of repetitions in the 30-seconds sit-to-stand test | At baseline, week 6, week 12, month 6 and month 9
  Changes in the number of repetitions in the 30-seconds sit-to-stand test
Changes in the score of the lower extremity functional scale | At baseline, week 12, month 6 and month 9
  Changes in the score of the lower extremity functional scale (LEFS). The LEFS is an 80-point questionnaire with 20 items scored from 0 to 4. A score of 80 means no disfunction while a score of 0 means maximal disfunction.
Changes in the score of the myotonic dystrophy health index | At baseline, week 6, week 12, month 6 and month 9
  Changes in the score of the myotonic dystrophy health index (MDHI). The MDHI is a 114-item questionnaire scored from 0 to 100, where 0 means no disability and 100 means maximal disability.
Changes in the score of the Fatigue and Daytime Sleepiness Scale | At baseline, week 6, week 12, month 6 and month 9
  Changes in the score of the Fatigue and Daytime Sleepiness Scale (FDSS). The FDSS is a 12-item questionnaire where all questions are scored from 0 to 2. A higher score means more daytime sleepiness and fatigue.
Changes in the Marin apathy scale | At baseline, week 12, month 6 and month 9
  Changes in the Marin apathy scale. The Marin apathy scale is scored by the clinician where he interviews the subject and then scores an 18-item list on a scale of 1 to 4. A high score means more apathy.
Changes in the Hospital Anxiety and Depression Scale | At baseline, week 6, week 12 and month 6
  Changes in the Hospital Anxiety and Depression Scale (HADS). The HADS is a 14-item questionnaire with a scale from 0 to 3 for each item. A high score means high depression and anxiety.
Changes in muscle biopsy of the vastus lateralis: muscle fiber typing | At baseline and week 12
  Changes in muscle biopsy of the vastus lateralis: muscle fiber typing
Changes in muscle biopsy of the vastus lateralis: muscle fiber size | At baseline and week 12
  Changes in muscle biopsy of the vastus lateralis: muscle fiber size (smallest diameter of the fiber)
Changes in muscle biopsy of the vastus lateralis: muscle proteomics | At baseline and week 12
  Changes in muscle biopsy of the vastus lateralis: muscle proteomics (protein expression)
Changes in muscle biopsy of the vastus lateralis: muscle transcriptomics | At baseline and week 12
  Changes in muscle biopsy of the vastus lateralis: muscle transcriptomics (RNA expression analysis)
Changes in muscle biopsy of the vastus lateralis: mitochondrial function | At baseline and week 12
  Changes in muscle biopsy of the vastus lateralis: mitochondrial function. Analysis of mitochondrial markers and enzymes
Changes in muscle biopsy of the vastus lateralis: Nuclear foci | At baseline and week 12
  Changes in muscle biopsy of the vastus lateralis: Nuclear foci (changes in accumulation of nuclear foci)
Changes in the time to perform of the Timed Up and Go | At baseline, week 6, week 12, month 6 and month 9
  Changes in the time to perform of the Timed Up and Go
Changes in the time to perform the Timed stair test | At baseline, week 6, week 12, month 6 and month 9
  Changes in the time to perform the Timed stair test
Change in the score of the Brief Pain Inventory | At baseline, week 6, week 12, month 6 and month 9
  Change in the score of the Brief Pain Inventory. The Brief Pain Inventory is a self-administer test that asses the dimensions of pain such as intensity of pain, functional incapacities, social and family repercussions, and psychological distress.
Self-perceived changes in daily life | At week 12
  Self-perceived changes in daily life
Change in the number of falls | At baseline, week 12, month 6 ans month 9
  Number of falls in the last week and in the last month
Change in score of the DM1-Activ questionnaire | At baseline, week 6, week 12, month 6 ans month 9
  Change in score of the DM1-Activ questionnaire. This questionnaire asses activity and social participation with DM1 population. It contains 20 items with a maximal socre of 40 points, a lower score represent a bigger impact of the disease on activities and social participation.
Change in blood : biochemical markers (CK, Protein C reactive, leukocytes, cytokines, etc.) | At baseline and week 12
  Change in blood : biochemical markers (CK, Protein C reactive, leukocytes, cytokines, etc.)
Change in urine sample : exercise biomarkers (-Omics markers) | At baseline and week 12
  Change in urine sample : exercise biomarkers (-Omics markers)
Change in saliva sample : exercise biomarkers (-Omics markers) | At baseline and week 12
  Change in saliva sample : exercise biomarkers (-Omics markers)
Change of the center of pressure (COP) measure in static posturography : open eyes bipodal position | At baseline, week 6, week 12, 6 months and 9 months
  Change of the center of pressure (COP) in static posturography : open eyes bipodal position
Change of the center of pressure (COP) measure in static posturography : closed eyes bipodal position | At baseline, week 6, week 12, 6 months and 9 months
  Change of the center of pressure (COP) in static posturography : closed eyes bipodal position
Change of the center of pressure (COP) measure in static posturography : open eyes semi-tandem position | At baseline, week 6, week 12, 6 months and 9 months
  Change of the center of pressure (COP) in static posturography : open eyes semi-tandem position
Change of the center of pressure (COP) measure in static posturography : open eyes tandem position | At baseline, week 6, week 12, 6 months and 9 months
  Change of the center of pressure (COP) in static posturography : open eyes tandem position

CONTACTS AND LOCATIONS:
Overall Officials: Elise Duchesne, Ph.D, Principal Investigator — Université du Québec à Chicoutimi
Locations (1):
- Groupe de recherche interdisciplinaire sur les maladies neuromusculaires, Saguenay, Quebec, Canada